CLINICAL TRIAL: NCT01751386
Title: A Double-Blind, Placebo-Controlled, Randomized Human Laboratory Pilot Study of Baclofen in Anxious Alcoholics
Brief Title: Baclofen for Treating Anxiety and Alcoholism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 130040; 13-AA-0040 (Other: The National Institutes of Health)
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-07-17

CONDITIONS: Alcoholism; Alcohol Dependence; Alcohol Drinking Related Problems; Alcohol Drinking; Anxiety Disorder
Keywords: Addiction; Cue-Induced Craving; Craving; Anxiety; Alcohol Consumption
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Anxiety Disorders; Behavior, Addictive | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Baclofen (Experimental): Baclofen 10 mg t.i.d.
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator): Placebo t.i.d.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Baclofen
  Arms: Baclofen
Other: Placebo
  Arms: Placebo

SUMMARY:
Background:

- Baclofen is a drug used to control muscle stiffness in people with neurological diseases. Some studies suggest that baclofen may reduce alcohol craving and use. It helps to reduce anxiety in alcoholics, which in turn can help to reduce cravings. Researchers want to see if baclofen can be a safe and effective treatment for alcoholics who have high anxiety levels.

Objectives:

- To see if baclofen is safe and helpful for people who have alcoholism and high anxiety levels.

Eligibility:

* Individuals between 21 and 65 years of age who have been diagnosed with alcoholism and anxiety issues.
* Participants must not be taking anti-anxiety medication.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Tests of alcohol dependency and anxiety levels will also be given.
* Participants will be divided into two groups. One group will take baclofen. The other group will have a placebo.
* About 1 week after the screening visit, participants will have a study visit. They will answer questions about their behavior and mood. They will then start to take either baclofen or a placebo. Participants will take the study drug three times a day, every day.
* After 1 week on the study drug, participants will have an overnight stay at the National Institutes of Health. They will have blood tests and answer questions about mood and behavior. They will also have tests that involve choosing to drink alcohol and answering more questions about cravings.
* Participants will stop taking their study drug over a 3-day period.
* A final follow-up visit will be required 1 week after the overnight study visit. Participants will receive information about other alcohol abuse treatment programs.

DETAILED DESCRIPTION:
Objective:

The selective GABAB receptor agonist baclofen has been identified as a possible medication able to reduce alcohol craving and intake in alcohol dependent individuals. In keeping with several preclinical studies, most of the clinical studies have demonstrated baclofen s effects in reducing alcohol craving and intake and promoting alcohol abstinence. However, one trial with alcoholics with a low severity of dependence found a robust treatment effect, but no differences between baclofen and placebo. The inconsistency of baclofen s effects on alcohol drinking among previous treatment trials suggests that different AD individuals may respond differently to baclofen. Baclofen has been demonstrated to consistently reduce anxiety in alcoholic patients, and analyses of positive vs. null findings with baclofen suggest that alcoholic patients with higher levels of anxiety at baseline may represent a sub-population particularly responsive to baclofen treatment. Therefore, this study will systematically test, for the first time, the specific role of baclofen on alcohol-related outcomes in alcoholic individuals with high anxiety levels. Furthermore, the biobehavioral mechanisms by which baclofen reduces drinking are not well characterized. A human laboratory pilot study conducted at Brown University with non-treatment seeking alcohol-dependent individuals suggests that baclofen reduces alcohol consumption both in the naturalistic environment as well as in a well-controlled lab setting (using an alcohol self-administration [ASA] paradigm) and that this could be mediated by baclofen s ability to alter alcohol-related biphasic effects. An exploratory analysis also revealed that specific genetic polymorphisms might moderate baclofen s effects, i.e. DRD4 and 5HTTLPR polymorphisms, although the sample of that pilot study was very small to allow one to draft definitive conclusions. The present project proposes investigating baclofen using a design similar to that used in the previous pilot study (thus, an already validated paradigm), thus representing not only the first study testing baclofen in alcoholic individuals with high anxiety levels, but also the first study investigating baclofen s biobehavioral mechanisms in such a population for which baclofen may hypothetically show a very robust effect.

Study population:

Non-treatment seeking alcohol-dependent males and females with high anxiety levels.

Design:

The experimental design is a between-subject randomized double-blind controlled study. The medication conditions baclofen t.i.d. or placebo represent the between subjects factor. Each participant will be randomly assigned to one of the two medication conditions and will receive eight days of the medication, followed by an alcohol laboratory session on Day 8. The alcohol laboratory session will be conducted in a bar-like room in the NIAAA Outpatient Clinic of the NIH CRC. The study will be conducted in consecutive phases which will appear contiguous to volunteers: (1) a one-week screening period; (2) an 8-day period (+ 1-5 days if needed to permit some participants flexibility in scheduling the laboratory session) during which participants will take the study medication; (3) an alcohol laboratory session, including a cue reactivity (CR) test and an alcohol self-administration (ASA) procedure on Day 8 (last day at the target dose); (4) a 3-day period during which participants will undergo a dose reduction of the study medication; (5) a 1-week follow-up (including the tapering phase).

Outcome measures:

Alcohol drinking during the ASA will be measured as the primary outcome. Secondary objectives include baclofen s effects on alcohol cue-induced responses (urge to drink, attention to cues, blood pressure, heart rate, saliva), on the subjective effects of alcohol and on anxiety levels. We will also explore the role of possible moderators of baclofen s effects, namely family history of alcoholism, early vs. later onset of alcoholism, pre-treatment anxiety levels and genetic moderators (DRD4, 5-HTTPRL). This study does not offer direct benefit to participants but is likely to yield generalizable knowledge about the possible role of baclofen in treating alcoholic individuals with high anxiety levels. This will markedly facilitate the identification of a novel pharmacotherapy, thus facilitating the development of novel alcoholism treatments.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must be male or female between 21 and 65 years old (inclusive).
* Participants must meet criteria for current DSM-IV-TR diagnosis of alcohol dependence, supported by the Structured Clinical Interview for DSM-IV-TR Axis I Disorders (SCID).
* Participants must have a Trait STAI > 39.
* Participants must be in good health as confirmed by medical history, physical examination, ECG, blood/urine lab tests.
* Females must be postmenopausal for at least one year, surgically sterile, or practicing an effective method of birth control before entry and throughout the study; have a negative urine pregnancy test at each visit. Reliable methods of birth control include oral contraceptives or Norplant ; barrier methods such as diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms with contraceptive foam, or intrauterine devices; a partner with a vasectomy; or abstinence from intercourse.

EXCLUSION CRITERIA:

* Individuals expressing interest in treatment for alcoholism and/or anxiety.
* Pregnancy or breast feeding women or not using an adequate form of birth control
* Unable to provide a negative urine drug screen.
* Individuals diagnosed with a current substance dependence diagnosis, other than alcohol or nicotine.
* Meet DSM-IV Axis I criteria for a lifetime diagnosis of schizophrenia, bipolar disorder, or other psychoses.
* An active illness within the past 6 months of Visit 1 that meet the DSM-IV criteria for a diagnosis of Major Depressive Disorder (MDD). Subjects with a history of attempted suicide will be excluded.
* Clinically significant medical abnormalities (i.e., unstable hypertension, clinically significant ECG abnormalities, Creatinine greater than or equal to 2 mg/dL). Although baclofen has demonstrated a safe profile when administered to alcoholic individuals with liver cirrhosis, including those with Hepatitis C, this study employs the oral administration of alcohol. Therefore, individuals with clinically significant liver problems will be excluded, i.e. liver cirrhosis, AST or ALT > 5 times the upper normal limit (UNL), and individuals with Hepatitis B and C.
* Current use of psychotropic medications that cannot be discontinued and that may have an effect on alcohol consumption (thus confounding the results of the study) or that may interact with baclofen. Specifically, contraindicated medications will include: naltrexone, acamprosate, alcohol dehydrogenase inhibitors, topiramate, gabapentin, ondansetron, benzodiazepines, beta-blockers, H2-blockers, and alpha-1 blockers.
* Medical contraindications for use of baclofen.
* A history of adverse reaction or hypersensitivity to baclofen.
* Participants who have significant alcohol withdrawal symptoms, defined as a CIWA-Ar > 8.
* History of epilepsy or alcohol-related seizures.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-12-03; Primary Completion 2016-08-17 (Actual); Study Completion 2016-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The NIH Biomedical Translational Research Information System

REFERENCES:
- [Background] Addolorato G, Abenavoli L, Leggio L, Gasbarrini G. How many cravings? Pharmacological aspects of craving treatment in alcohol addiction: a review. Neuropsychobiology. 2005;51(2):59-66. doi: 10.1159/000084161. Epub 2005 Feb 28. PMID 15741745
- [Background] Addolorato G, Caputo F, Capristo E, Domenicali M, Bernardi M, Janiri L, Agabio R, Colombo G, Gessa GL, Gasbarrini G. Baclofen efficacy in reducing alcohol craving and intake: a preliminary double-blind randomized controlled study. Alcohol Alcohol. 2002 Sep-Oct;37(5):504-8. doi: 10.1093/alcalc/37.5.504. PMID 12217947
- [Background] Addolorato G, Caputo F, Capristo E, Janiri L, Bernardi M, Agabio R, Colombo G, Gessa GL, Gasbarrini G. Rapid suppression of alcohol withdrawal syndrome by baclofen. Am J Med. 2002 Feb 15;112(3):226-9. doi: 10.1016/s0002-9343(01)01088-9. No abstract available. PMID 11893350
- [Background] Leggio L, Zywiak WH, Edwards SM, Tidey JW, Swift RM, Kenna GA. A preliminary double-blind, placebo-controlled randomized study of baclofen effects in alcoholic smokers. Psychopharmacology (Berl). 2015 Jan;232(1):233-43. doi: 10.1007/s00213-014-3652-9. Epub 2014 Jun 29. PMID 24973894
- [Background] Leggio L, Zywiak WH, McGeary JE, Edwards S, Fricchione SR, Shoaff JR, Addolorato G, Swift RM, Kenna GA. A human laboratory pilot study with baclofen in alcoholic individuals. Pharmacol Biochem Behav. 2013 Feb;103(4):784-91. doi: 10.1016/j.pbb.2012.11.013. Epub 2012 Dec 19. PMID 23262301
- [Background] Leggio L, Ferrulli A, Zambon A, Caputo F, Kenna GA, Swift RM, Addolorato G. Baclofen promotes alcohol abstinence in alcohol dependent cirrhotic patients with hepatitis C virus (HCV) infection. Addict Behav. 2012 Apr;37(4):561-4. doi: 10.1016/j.addbeh.2011.12.010. Epub 2011 Dec 27. PMID 22244707
- [Result] Farokhnia M, Schwandt ML, Lee MR, Bollinger JW, Farinelli LA, Amodio JP, Sewell L, Lionetti TA, Spero DE, Leggio L. Biobehavioral effects of baclofen in anxious alcohol-dependent individuals: a randomized, double-blind, placebo-controlled, laboratory study. Transl Psychiatry. 2017 Apr 25;7(4):e1108. doi: 10.1038/tp.2017.71. PMID 28440812
- [Derived] Richardson RS, Farokhnia M, Vendruscolo LF, Leggio L. Plasma concentrations of the inflammatory adipokine lipocalin-2 are not affected by chronic alcohol exposure in rats or acute alcohol administration in people with alcohol use disorder. Am J Drug Alcohol Abuse. 2025;51(6):730-740. doi: 10.1080/00952990.2025.2582563. Epub 2025 Dec 2. PMID 41329966
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-AA-0040.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Baclofen: Baclofen capsules: 15 mg/day (5 mg t.i.d.; titration phase) for 3 days, followed by 30 mg/day (10 mg t.i.d.; target dose) until the alcohol laboratory session; then, 15 mg/day (5 mg t.i.d.; taper down) for three additional days.
- Placebo: Placebo capsules, similar to baclofen in appearance, texture, taste, and odor
Period: Overall Study
Arm/Group | Baclofen | Placebo
Started | 20 | 19
Completed | 18 | 16
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baclofen | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 6 | 4 | 10
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Alcohol Consumed During the Alcohol Self Administration (ASA) Session
Description: Amount of alcohol was measured as the number of mini-drinks each participant decided to drink (0-8 mini-drinks). The alcohol content of each mini-drink was calculated based on the participants' total body water, and was designed to raise the blood alcohol concentration by 0.015 g/dL.
Time Frame: 2 hours
Population: The analysis included all subjects who took the medication (either baclofen or placebo) and finished the alcohol laboratory session
Measure: Mean (Standard Error); unit: mini-drinks
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 18 | 16
mini-drinks | 4.11 (0.66) | 4.5 (0.72)

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Baclofen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 9/20 | 7/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Baclofen (N=20) | Placebo (N=19)
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Decreased appetite (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 3
Insomnia (Nervous system disorders) | 3 | 2
Memory impairment (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 4 | 5
Depression (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes